CLINICAL TRIAL: NCT02707497
Title: The Effect of Recombinant Human Thrombopoietin(rhTPO) on Sepsis Patients With Acute Severe Thrombocytopenia：a Prospective, Multi-center, Open-label, ,Randomized, Controlled Trial
Brief Title: The Effect of REcombinant Human Thrombopoietin (rhTPO) on Sepsis Patients With aCUte Severe thrombocytopEnia
Acronym: RESCUE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ruilan Wang (Other)
Collaborators: Huadong Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Changhai Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Shanghai Jiao Tong University School of Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); Fudan University (Other)
Responsible Party: Sponsor-Investigator, Ruilan Wang, The director of emergency and intensive care unit, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RWang-TPO-301
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Sepsis; Thrombocytopenia
Keywords: sepsis; severe thrombocytopenia; recombinant human thrombopoietin; platelets; 28-day mortality
MeSH Terms: conditions — Sepsis; Thrombocytopenia | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTPO (Experimental): Recombinant Human Thrombopoietin，TPIAO®, Shenyang Sunshine Pharmaceutical Company Limited [SUNSHINE], Shenyang, China）， 15000u/d, qd, subcutaneous injection, daily for no more than 7 consecutive days
  Interventions: Drug: rhTPO
- placebo (Placebo Comparator): The control group will not use any platelet-increased drugs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhTPO — Recombinant Human Thrombopoietin，TPIAO®, Shenyang Sunshine Pharmaceutical Company Limited [SUNSHINE], Shenyang, China）， 15000u/d, qd, subcutaneous injection, daily for no more than 7 consecutive days
  Other Names: Recombinant Human TPO
  Arms: rhTPO
Drug: Placebo — The control group will not use any platelet-increased drugs.
  Other Names: No platelet-increased drug
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether recombinant human thrombopoietin(rhTPO) can rapidly increase the platelets counts, shorten the time of the platelet returned to normal, reduce platelet transfusion and bleeding events, prompt recovery of organ function, decrease the length of ICU stay, and eventually reduce the 28-day mortality in sepsis patients with severe thrombocytopenia.

DETAILED DESCRIPTION:
Sepsis is a high morbidity and mortality in critical care unit. Clinically, we found that secondary thrombocytopenia was common in the patients with sepsis, and the incidence can be as high as 55%. Moreover, many studies have shown that thrombocytopenia is an early prognostic marker in sepsis and an independent risk factor for the mortality of sepsis. Furthermore, sepsis patients with severe thrombocytopenia(PLT< 50×10^9/L) have the higher mortality of 50%-90%. And then, it has been reported that early recovery from thrombocytopenia helps to prevent the coagulopathy and decreases the mortality. Until now, the treatment of thrombocytopenia are mainly platelet transfusion and platelet-increased drugs. Because of source scarcity, transfusion-related infectious and immunological complications, platelet transfusion is limited in the clinical treatment. So, the use of platelet-increased drugs for replacement therapy becomes an inevitable trend. The primary purpose of this study is to explore the effect of platelet-increased drugs (rhTPO) on sepsis patients with severe thrombocytopenia.

The study is designed as a prospective, multi-center, open-label, randomized, controlled trial in 7 tertiary academic medical centers which are medical, surgical or general ICUs. Patient enrollment is expected to last up to 30 months. Eligible patients will be randomly assigned to the control and rhTPO add-on treatment in a dynamic random and competitive design in clinical trial sites. Sequential organ failure assessment (SOFA), Acute Physiology and Chronic Health Evaluation II (APACHE II) scores are as the dynamic equilibrium factors. Randomization will be done after the first assessment, ensuring that the assessing occupational therapist will not be biased at this time by knowing the group assignment. Both groups receive appropriate medical support and treatment based on guidelines issued by the surviving sepsis campaign.

The intervention group will receive rhTPO at a dose of 15000u/d, subcutaneous injection, for 7 consecutive days. It will be terminated when platelet counts (PCs) reach the standard of clinical recovery of platelets: increased by 50×10^9/L for 3 consecutive days compared with PCs at baseline, or PCs are more than 100×10^9/L, or the duration of rhTPO is more than 7 days. The time from randomization to administration of rhTPO will be within 24 hours. The control group will not use any platelet-increased drugs.

Platelet transfusion is advised to be administered when PCs are below 10×10^9/L in the absence of apparent bleeding; or below 20 ×10^9/L if the patient has a significant risk of bleeding in both two groups; or below 50 ×10^9/L if the patient has active bleeding or need invasive operation.

Patients will be followed for 28 days. PCs will be monitored every day until the first 7 days, followed by tests once a week. Liver and renal function, coagulation function, inflammatory biomarkers (CRP, PCT), and the severity of the disease (SOFA, APACHEǁ) will be monitored before treatment, followed by tests once a week. And then, the number of blood transfusion (including platelets), the length of ICU stay, days free from advanced cardiovascular/respiratory/renal support, bleeding events, and any adverse effects will be recorded after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed or clinical diagnosed infection
2. The change of Sequential Organ Failure Assessment(ΔSOFA) score ≥ 2
3. PLT< 50×10^9/L
4. Informed consent

Exclusion Criteria:

1. History of the treatments with chemotherapeutic drugs or heparin within six months
2. History of bone marrow stem cell disorders, malignancy, or immunologic diseases
3. History of bone marrow, lung, liver, kidney, pancreas, or small bowel transplantation.
4. Confirmed End-stage renal failure(GFR <10ml/min，Scr>707μmol/L)
5. Confirmed Disseminated Intravascular Coagulation(DIC)
6. Confirmed Hemorrhagic brain injury or need craniocerebral operation
7. Died anticipated within 24 hours
8. Known pregnancy or at breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days after enrolled
  The 28-day mortality of the patients

SECONDARY OUTCOMES:
The changes of platelets counts (PCs) in the first 7 days | 7 days after enrolled
  The changes of PCs in the first 7 days
The clinical recovery time of PCs | 28 days after enrolled
  The time of PCs that reach the standard of clinical recovery
The amount of blood transfusion | 28 days after enrolled
  The amount of blood transfusion (including platelets, RBC, FP)
The proportion of blood transfusion | 28 days after enrolled
  The proportion of patients who need blood transfusion(including platelets, RBC, FP)
The changes of procalcitonin | 28 days after enrolled
  The data of procalcitonin (PCT) in different time points
The changes of C-reactive protein | 28 days after enrolled
  The data of C-reactive protein (CRP) in different time points
The changes of endotoxin | 28 days after enrolled
  The data of endotoxin in different time points
The changes of D-dimer and Fibrinogen | 28 days after enrolled
  The data of D-dimer and Fibrinogen in different time points
The changes of PT and APTT | 28 days after enrolled
  The data of PT and APTT in different time points
The changes of liver function | 28 days after enrolled
  The data of the markers of liver function (including ALT, AST, TBIL, DBIL) in different time points
The changes of renal function | 28 days after enrolled
  The data of the markers of renal function (including serum Cr and BUN) in different time points
The changes of cardiac function | 28 days after enrolled
  The data of the markers of cardiac function (including Troponin I and BNP) in different time points
The days free from advanced organ support | 28 days after enrolled
  The days without advanced cardiovascular/respiratory/ renal support within 28 days
The incidence of bleeding event | 28 days after enrolled
  The incidence of bleeding event, according to Bleeding Academic Research Consortium Definition for Bleeding
The incidences of drug-related adverse events | 28 days after enrolled
  The incidences of drug-related adverse events as assessed by CTCAE v4.0
The length of ICU and hospital stay | 28 days after enrolled
  The days from enrolled to discharge from ICU or hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ruilan Wang, MD,PhD, Principal Investigator — The department of ICU, Shanghai General Hospital, Shanghai Jiaotong University
Locations (1):
- Shanghai General Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication.

REFERENCES:
- [Derived] Zhou Z, Feng T, Xie Y, Huang P, Xie H, Tian R, Qian B, Wang R. The effect of recombinant human thrombopoietin (rhTPO) on sepsis patients with acute severe thrombocytopenia: a study protocol for a multicentre randomised controlled trial (RESCUE trial). BMC Infect Dis. 2019 Sep 6;19(1):780. doi: 10.1186/s12879-019-4388-2. PMID 31492102